CLINICAL TRIAL: NCT03234400
Title: A Phase 1, Randomized Pharmacokinetics and Safety Study of Extended Duration Dapivirine Vaginal Rings
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MTN-036/IPM 047; 5UM1AI068633 (NIH)
Record Dates: First submitted 2017-07-25; First posted 2017-07-31 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- 25 mg Dapivirine Vaginal Ring (Experimental): Participants will insert one Dapivirine Vaginal Ring, 25 mg to be replaced every 4 weeks for 8 weeks, then worn for an additional 5 weeks for a total of 13 weeks. Participants will continue follow-up for an additional one to three days after final VR removal.
  Interventions: Combination Product: Dapivirine Vaginal Ring, 25 mg
- 100 mg Dapivirine Vaginal Ring (Experimental): Participants will insert one Dapivirine Vaginal Ring, 100 mg to be used continuously for 13 weeks. Participants will continue follow-up for an additional one to three days after final VR removal.
  Interventions: Combination Product: Dapivirine Vaginal Ring, 100 mg
- 200 mg Dapivirine Vaginal Ring (Experimental): Participants will insert one Dapivirine Vaginal Ring, 200 mg to be used continuously for 13 weeks. Participants will continue follow-up for an additional one to three days after final VR removal.
  Interventions: Combination Product: Dapivirine Vaginal Ring, 200 mg

INTERVENTIONS:
Combination Product: Dapivirine Vaginal Ring, 25 mg — Vaginal Ring containing 25 mg dapivirine
  Arms: 25 mg Dapivirine Vaginal Ring
Combination Product: Dapivirine Vaginal Ring, 100 mg — Vaginal Ring containing 100 mg dapivirine
  Arms: 100 mg Dapivirine Vaginal Ring
Combination Product: Dapivirine Vaginal Ring, 200 mg — Vaginal Ring containing 200 mg dapivirine
  Arms: 200 mg Dapivirine Vaginal Ring

SUMMARY:
Participants will be randomized to one of three study vaginal rings (VRs) in a 1:1:1 ratio, 25 mg, 100 mg or 200 mg VRs.

DETAILED DESCRIPTION:
Participants will be randomized to one of three study vaginal rings (VRs) in a 1:1:1 ratio, and those randomized to the 100 mg and 200 mg VRs will not be told their group assignment. Participants will insert one VR to be used continuously for 13 weeks (100 mg VR or 200 mg VR) or one VR (25 mg VR) to be replaced every 4 weeks for 8 weeks, then worn for an additional 5 weeks for a total of 13 weeks. Participants will continue follow-up for an additional one to three days after final VR removal.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female sex at birth Note: Participants who are female at birth, who now identify as male, will not be excluded so long as they are not on female-to-male transition therapy.
* Age 18 through 45 years (inclusive) at Screening, verified per site SOPs
* Able and willing to provide written informed consent to be screened for and enrolled in MTN-036/IPM 047
* Able and willing to provide adequate locator information, as defined in site SOPs
* Able to communicate in spoken and written English
* Available for all visits and able and willing to comply with all study procedural requirements
* Willing to comply with abstinence and other protocol requirements
* Willing to use male condoms for penile-vaginal intercourse (PVI) and penile-rectal intercourse for the duration of study participation
* Per participant report, using an effective method of contraception for at least 30 days (inclusive) prior to Enrollment, and intending to continue use of an effective method for the duration of study participation; effective methods include:

  1. hormonal methods (except contraceptive ring)
  2. intrauterine device (IUD)
  3. sterilization (of participant or partner, as defined in site SOPs)
  4. having sex exclusively with cis-women
  5. abstinence from PVI for 90 days prior to Enrollment, and intending to remain abstinent from PVI for the duration of study participation
* HIV-uninfected based on testing performed at Screening and Enrollment
* Per participant report at Screening, regular menstrual cycles with at least 21 days between menses Note: This criterion is not applicable to participants who report using a progestin-only method of contraception at Screening (e.g., Depo-Provera or levonorgestrel-releasing IUD) nor to participants using continuous combination oral contraceptive pills, as the absence of regular menstrual cycles is an expected, normal consequence in this context.
* Per participant report at Screening and Enrollment, states a willingness to refrain from inserting any non-study vaginal products or objects into the vagina including, but not limited to spermicides, female condoms, diaphragms, intravaginal rings, vaginal medications, menstrual cups, cervical caps, douches, lubricants, and sex toys (vibrators, dildos, etc.) for the 24 hours preceding the Enrollment Visit and for the duration of study participation.

Note: Use of tampons is permitted except for 24 hours prior to clinic visits in which CVF samples are scheduled to be collected.

* Participants over the age of 21 (inclusive) must have documentation of a satisfactory Pap within the past 3 years prior to Enrollment consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 (Dated November 2007) to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Version 2.1, March 2017, or satisfactory evaluation with no treatment required of Grade 1 or higher Pap result
* At Screening and Enrollment, agrees not to participate in other research studies involving drugs, medical devices, vaginal products or vaccines after the Screening Visit and for the duration of study participation

Exclusion Criteria:

* Pregnant at Screening or Enrollment or plans to become pregnant during the study period
* Diagnosed with a UTI or reproductive tract infection (RTI) at Screening or Enrollment
* Diagnosed with an acute STI requiring treatment per current Centers for Disease Control and Prevention (CDC) guidelines (http://www.cdc.gov/std/treatment/) at Screening or Enrollment such as gonorrhea (GC), CT, trichomonas, PID, and/or syphilis
* Has a clinically apparent Grade 2 or higher pelvic exam finding (observed by study staff) at Screening or Enrollment, as per the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1, March 2017, and/or Addendum 1 (Female Genital Grading Table for Use in Microbicide Studies [Dated November 2007])
* 5) Participant report and/or clinical evidence of any of the following:

  1. Known adverse reaction to any of the study products (ever)
  2. Chronic and/or recurrent vaginal candidiasis
  3. Non-therapeutic injection drug use in the 12 months prior to Enrollment
  4. Last pregnancy outcome less than 90 days prior to Enrollment
  5. Gynecologic or genital procedure (e.g., tubal ligation, dilation and curettage, piercing) 45 days or less prior to Enrollment Note: Colposcopy and cervical biopsies for evaluation of an abnormal Pap test as well as IUD insertion/removal are not exclusionary.
  6. Currently breastfeeding or planning to breastfeed during the study period
  7. Participation in any other research study involving drugs, medical devices, vaginal products or vaccines, in the 60 days prior to Enrollment
* Use of pre-exposure prophylaxis (PrEP) for HIV prevention and/or post-exposure prophylaxis (PEP) for potential HIV exposure within the 3 months prior to Enrollment, and/or anticipated use and/or unwillingness to abstain from PrEP during trial participation
* Has any of the following Grade 1 or higher laboratory abnormalities at Screening Visit:

  1. AST or ALT
  2. Hemoglobin
* Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate the interpretation of study outcome data, or otherwise interfere with achieving the study objectives including any significant uncontrolled active or chronic medical condition.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
DPV concentration in plasma. | 13 weeks
  To compare the local and systemic pharmacokinetics (PK) of two extended duration DPV VRs (100 mg and 200 mg) when used continuously for 13 weeks to the current 25 mg DPV VR when replaced every 4 weeks for 8 weeks and then worn for an additional 5 weeks for a total of 13 weeks.
DPV concentration in cervicovaginal fluid | 13 weeks
  To compare the local and systemic pharmacokinetics (PK) of two extended duration DPV VRs (100 mg and 200 mg) when used continuously for 13 weeks to the current 25 mg DPV VR when replaced every 4 weeks for 8 weeks and then worn for an additional 5 weeks for a total of 13 weeks.
DPV concentration in cervical tissue | 13 weeks
  To compare the local and systemic pharmacokinetics (PK) of two extended duration DPV VRs (100 mg and 200 mg) when used continuously for 13 weeks to the current 25 mg DPV VR when replaced every 4 weeks for 8 weeks and then worn for an additional 5 weeks for a total of 13 weeks.
Safety comparison of the two extended duration DPV VRs (100 mg and 200 mg) to the current 25 mg DPV VR | 13 weeks
  * Proportions of participants with Grade 2 or higher genitourinary adverse events as defined by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1, March 2017, and/or Addendum 1 (Female Genital Grading Table for Use in Microbicide Studies [Dated November 2007])
  * Proportions of participants with Grade 3 or higher adverse events as defined by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1, March 2017

SECONDARY OUTCOMES:
Adherence | 13 weeks
  • Frequency of study VR removal/expulsions (voluntary and involuntary) and duration without VR in vagina (by self-report)
Adherence | 13 weeks
  • VR use initiation and persistence (whether the VR is in place when participants come to the clinic for their study visits)
Acceptability | 13 weeks
  Degree to which study participants liked or disliked using the three DPV VRs (by self-report)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Bridge HIV CRS San Francisco Department of Public Health, San Francisco, California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hawley I, Song M, Scheckter R, McClure T, Piper J, Chen BA, Hoesley C, Liu AY, van der Straten A. Users' Preferred Characteristics of Vaginal Rings for HIV Prevention: A Qualitative Analysis of Two Phase I Trials. AIDS Res Hum Retroviruses. 2022 Apr;38(4):313-326. doi: 10.1089/AID.2021.0077. Epub 2022 Feb 11. PMID 34969254
- [Derived] Liu AY, Dominguez Islas C, Gundacker H, Neradilek B, Hoesley C, van der Straten A, Hendrix CW, Beamer M, Jacobson CE, McClure T, Harrell T, Bunge K, Devlin B, Nuttall J, Spence P, Steytler J, Piper JM, Marzinke MA; MTN-036/IPM 047 Protocol Team for the Microbicide Trials Network. Phase 1 pharmacokinetics and safety study of extended duration dapivirine vaginal rings in the United States. J Int AIDS Soc. 2021 Jun;24(6):e25747. doi: 10.1002/jia2.25747. PMID 34118115